CLINICAL TRIAL: NCT03083171
Title: A Randomized Double-blind Placebo-controlled Phase I Study on the Safety, Tolerability and Pharmacokinetics/-Dynamics of Escalating Single Intravenous Doses of ADRECIZUMAB (HAM8101) in Healthy Male Subjects During Experimental Endotoxemia.
Brief Title: Adrecizumab-LPS Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adrenomed AG (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Adrecizumab-LPS
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: Adrecizumab; Adrenomedullin; Healthy volunteers; LPS; Monoclonal recombinant antibody
MeSH Terms: interventions — Endotoxins; Lipopolysaccharides; enibarcimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Endotoxin; Drug: Placebo
- Adrecizumab 0.5 mg/kg (Active Comparator): A single intravenous dose of 0.5 mg/kg Adrecizumab given over a 1 hour period.
  Interventions: Drug: Endotoxin; Drug: Adrecizumab
- Adrecizumab 2.0 mg/kg (Active Comparator): A single intravenous dose of 2.0 mg/kg Adrecizumab given over a 1 hour period.
  Interventions: Drug: Endotoxin; Drug: Adrecizumab
- Adrecizumab 8.0 mg/kg (Active Comparator): A single intravenous dose of 8.0 mg/kg Adrecizumab given over a 1 hour period.
  Interventions: Drug: Endotoxin; Drug: Adrecizumab

INTERVENTIONS:
Drug: Endotoxin — At T=0 1 ng/kg E. Coli type O113 lipopolysaccharide is administrated intravenously as a bolus, followed by 1 ng/kg/hour for 3 hours.
  Other Names: LPS; Lipopolysaccharide
Drug: Placebo — At T=1 hour, placebo will be administered intravenously over a 1 hour period. Placebo is indistinguishable from Adrecizumab.
  Arms: Placebo
Drug: Adrecizumab — At T=1 hour, Adrecizumab will be administered intravenously over a 1 hour period.
  Arms: Adrecizumab 0.5 mg/kg; Adrecizumab 2.0 mg/kg; Adrecizumab 8.0 mg/kg

SUMMARY:
In this randomized, double-blind, placebo-controlled study, either a single dose of Adrecizumab (0.5, 2.0 or 8.0 mg/kg) or placebo will be administrated to 24 healthy male volunteers during experimental endotoxemia.

DETAILED DESCRIPTION:
Adrenomedullin (ADM) is a natural occurring 52 amino acid peptide which is mainly expressed in endothelial and smooth muscle cells. ADM plasma levels are increased in patients with sepsis and related with severity of disease. ADM is a key regulator of vasotonus and of endothelial integrity in sepsis. Adrecizumab is an antibody against the N-terminus of ADM which only partially inhibits the bioactivity of ADM. Several septic animal studies have shown that administration of Adrecizumab leads to stabilization of hemodynamics in mice and pigs, improved renal function, reduced catecholamine demand, improved fluid balance and improved survival. The administration of Adrecizumab to rodents, non-human primates and recently humans, has been tolerated very well.

The experimental human endotoxemia model, in which healthy male volunteers receive a low dose of lipopolysaccharide (LPS) derived from Escherichia coli, is widely used to study the effects of systemic inflammation in humans in vivo and is considered a safe and highly reproducible method to activate the innate immune system. Furthermore, previous data has shown that experimental human endotoxemia results in increased plasma ADM levels. In this study, the investigators wish to assess the safety, tolerability and pharmacokinetics/-dynamics of Adrecizumab under inflammatory conditions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in this trial prior to any study-mandated procedure.
2. Male subjects aged 18 to 35 years inclusive.
3. Subjects have to agree to use a reliable way of contraception with their partners from study entry until 3 months after study drug administration.
4. BMI between 18 and 30 kg/m², with a lower limit of body weight of 50 kg and a upper limit of 100 kg.
5. Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory parameters.

Exclusion Criteria:

1. Unwillingness to abstain from any medication, including recreational drugs or vitamin supplements during the course of the study and within 7 days prior to the treatment day.
2. Unwillingness to abstain from smoking, or alcohol, within 1 day prior to the treatment day and 1 day after the treatment day.
3. Previous participation in a trial where LPS was administered.
4. Surgery or trauma with significant blood loss or blood donation within 3 months prior to the treatment day.
5. History, signs or symptoms of cardiovascular disease, in particular:

   * History of frequent vasovagal collapse or of orthostatic hypotension
   * Resting pulse rate ≤45 or ≥100 beats/min
   * Hypertension (RR systolic >160 or RR diastolic >90 mmHg)
   * Hypotension (RR systolic <100 or RR diastolic <50 mmHg)
   * Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
   * Any chronic cardiac arrhythmias (except PAC's, PVC's)
6. Renal impairment: plasma creatinine >120 μmol/L
7. Liver function tests (alkaline phosphatase, AST, ALT and/or γ-GT) above 2x the upper limit of normal.
8. History of asthma
9. Atopic constitution
10. CRP above 2x the upper limit of normal, or clinically significant acute illness, including infections, within 2 weeks prior to the treatment day.
11. Treatment with investigational drugs or participation in any other clinical trial within 30 days prior to the treatment day.
12. Known or suspected of not being able to comply with the trial protocol.
13. Known hypersensitivity to any excipients of the drug formulations used.
14. Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability expressed in total number of treatment related (serious) adverse events. | 3 months follow-up period
  Adverse events include: Clinically significant variation in vital signs compared to baseline (blood pressure and heart rate), local infusion reaction at site of i.v. IMP infusion, clinically significant changes in ECG compared to baseline and clinically significant deflections in laboratory parameters compared to baseline.

SECONDARY OUTCOMES:
Area under the curve (AUC) of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days after Adrecizumab administration
Peak plasma concentration (Cmax) of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days after Adrecizumab administration
Terminal t1/2 of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days after Adrecizumab administration
Clearance of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days after Adrecizumab administration
Volume of distribution of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days after Adrecizumab administration
Plasma levels of adrenomedullin and MR-proadrenomedullin | T=0 hours, T=1 hours, T=1.25 hours, T=1.5 hours, T=2 hours, T=2.5 hours T=3 hours, T=4 hours, T=5 hours, T=9 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days after LPS administration
Cytokines | T=0 hours, T=1 hours, T=1.5 hours, T=2 hours, T=2.5 hours T=3 hours, T=4 hours, T=5 hours, T=6 hours, T=9 hours after LPS administration
  Blood plasma levels of TNF-alfa, IL-6, IL-8, IL-10, MCP-1, IP-10 and G-CSF
Kidney damage markers | Baseline, T=0 to T=3 hours, T=3 to T=6 hours, T=6 to T=9 hours, T=9 to T=12 hours, T=12 to T=24 hours after LPS administration
  In urine and plasma, including, but not limited to pro-enkephalin, creatinine clearance, NGAL and KIM-1

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Dept. of Intensive Care Medicine, Research-unit, Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided